CLINICAL TRIAL: NCT02183363
Title: Bioavailability of BI 1356 After Single Oral Administration of 5 mg BI 1356 Given as Tablet Formulation TF IIb Relative to Tablet Formulation TF II and Tablet Formulation iFF in Healthy Male Volunteers (an Open Label, Randomised, Single-dose, Three-way Crossover Study)
Brief Title: Bioavailability of BI 1356 After Single Oral Administration Given as Different Tablet Formulation in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.25
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- BI 1356 - Tablet TFII (Experimental)
  Interventions: Drug: BI 1356 - Tablet TFII; Drug: BI 1356 - Tablet iFF; Drug: BI 1356 - Tablet TFIIb
- BI 1356 - Tablet iFF (Experimental)
  Interventions: Drug: BI 1356 - Tablet TFII; Drug: BI 1356 - Tablet iFF; Drug: BI 1356 - Tablet TFIIb
- BI 1356 - Tablet TFIIb (Active Comparator)
  Interventions: Drug: BI 1356 - Tablet TFII; Drug: BI 1356 - Tablet iFF; Drug: BI 1356 - Tablet TFIIb

INTERVENTIONS:
Drug: BI 1356 - Tablet TFII
Drug: BI 1356 - Tablet iFF
Drug: BI 1356 - Tablet TFIIb

SUMMARY:
Study to investigate the relative bioavailability of 5 mg BI 1356 as tablet formulations (Trial formulation) TF II and Intended final formulation (iFF) vs. 5 mg BI 1356 as tablet TF IIb

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs, Blood Pressure (BP), Pulse Rate (PR), 12-lead Electrocardiogram (ECG), clinical laboratory tests

  * No findings deviating from normal and of clinical relevance
  * No evidence of a clinically relevant concomitant disease
* Age ≥21 and Age ≤55 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
AUC0-24 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours) | predose, up to 24 hours

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | predose, up to 264 hours
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | predose, up to 264 hours
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | predose, up to 264 hours
AUCt1-t2 (Partial area under the concentration time curve of the analyte in plasma over the time interval t1 to t2) | predose, up to 264 hours
C24 (plasma concentration of the analyte 24 hours after dosing) | predose, up to 264 hours
tmax (time from dosing to the maximum concentration of the analyte in plasma) | predose, up to 264 hours
λz (terminal rate constant in plasma) | predose, up to 264 hours
t1/2 (terminal half-life of the analyte in plasma) | predose, up to 264 hours
MRTpo (mean residence time of the analyte in the body after po administration) | predose, up to 264 hours
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | predose, up to 264 hours
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | predose, up to 264 hours
Changes in Dipeptidyl-peptidase-IV (DPP-IV) activity in plasma | predose, up to 264 hours
Changes in plasma glucose levels | predose, up to 264 hours
Number of patients with adverse events | up to 18 days following last drug administration
Number of patients with abnormal findings in physical examination | up to 18 days following last drug administration
Number of patients with clinically significant changes in vital signs (Blood Pressure (BP), Pulse Rate (PR)) | up to 18 days following last drug administration
Number of patients with abnormal changes 12-lead ECG (electrocardiogram) | up to 18 days following last drug administration
Number of patients with abnormal changes in laboratory parameters | up to 18 days following last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 18 days following last drug administration